CLINICAL TRIAL: NCT05387057
Title: Effectiveness of an Individualized Exergame-based Motor-Cognitive Training Concept Targeted to Improve Cognitive Functioning in Older Adults With Mild Neurocognitive Disorder - A Randomized Controlled Trial
Brief Title: Effectiveness of a Novel Exergame-Based Training Concept for Older Adults With Mild Neurocognitive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eling DeBruin (Other)
Responsible Party: Sponsor-Investigator, Eling DeBruin, Prof. Dr., Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BASEC Nr. 2022-00386
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Mild Neurocognitive Disorder
Keywords: Exergames; Mild Neurocognitive Disorder; Cognition; Neuroscience; Exercise; Training
MeSH Terms: conditions — Neurocognitive Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Allocation ratio = 1 (Intervention) : 1 (Control) stratified by gender and per institute (study site)
Who Masked: Outcomes Assessor
Masking Description: The study will be conducted as a single-blinded study: the outcome evaluator of the pre- and post-measurements will be blinded to group allocation. Blinding of participants will not be possible since usual care will be used as a control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Exergame Training (Experimental): Participants in the intervention group will perform a twelve-week training intervention in addition to their usual care (as provided by the (memory) clinics where the patients are recruited). The training intervention will be prescribed according to our newly developed exergame-based training concept (called 'Brain-IT' exergame-based training concept). Our complete 'Brain-IT' exergame-based training concept has recently been published including sufficient details about the exergame components as well as the exercise and training characteristics (i.e. including all predefined levels of task demands as well as the detailed progression rules) to allow full replication (i.e. consider supplementary file 3 of doi: 10.3389/fnagi.2021.734012). This training concept was planned and will be reported using the Consensus on Exercise Reporting Template (CERT; doi: 10.1136/bjsports-2016-096651).
  Interventions: Behavioral: Exergame training according to the 'Brain-IT' exergame-based training concept
- Usual Care (Active Comparator): The control group will proceed with usual care as provided by the (memory) clinics where the patients are recruited.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Exergame training according to the 'Brain-IT' exergame-based training concept — For an overview, our 'Brain-IT' exergame-based training concept consists of an individually adapted multi-domain exergame-based simultaneous cognitive-motor training with incorporated cognitive tasks that will be adopted with a deficit-oriented focus on the neurocognitive domains of (1) learning and memory, (2) executive function, (3) complex attention, and (4) visuospatial skills. According to the training concept, each participant is instructed to train 5x/week for 24 min per session resulting in a weekly exercise volume of 120 min. All training sessions are planned to take place at participant's homes using the exergame training system 'Senso Flex' (Dividat AG, Schindellegi, Switzerland). For a detailed description of the complete 'Brain-IT' exergame-based training concept with sufficient details to allow full replication, consider our methodological paper (doi: 10.3389/fnagi.2021.734012).
  Arms: Intervention Group - Exergame Training
Behavioral: Usual Care — The control group will proceed with usual care as provided by the (memory) clinics where the patients are recruited.
  Arms: Usual Care

SUMMARY:
BACKGROUND:

Simultaneous motor-cognitive training interventions are considered promising to prevent the decline in cognitive functioning in older adults with mild neurocognitive disorder (mNCD) and can be highly motivating when applied in form of exergames.

OBJECTIVES:

This study systematically explores the effectiveness of a newly developed exergame-based motor-cognitive training concept (called 'Brain-IT') targeted to improve cognitive functioning in older adults with mNCD.

METHODS:

A two-arm, parallel-group, single-blinded (i.e. outcome evaluator of pre- and post-measurements blinded to group allocation) randomized controlled trial with an allocation ration of 1 : 1 (i.e. intervention : control) including 34 - 40 older adults with mNCD will be conducted between May 2022 and December 2023. The control group will proceed with usual care as provided by the (memory) clinics where the patients are recruited while the intervention group will perform a twelve-week training intervention according to the newly developed 'Brain-IT' exergame-based training concept in addition to usual care. As a primary outcome, global cognitive functioning will be assessed using the Quick Mild Cognitive Impairment Screen (Qmci). As secondary outcomes, domain-specific cognitive functioning, brain structure and function, spatiotemporal parameters of gait, instrumental activities of daily living, psychosocial factors (e.g. quality of life, and levels of depression, anxiety, stress), and cardiac vagal modulation (heart rate variability at rest) will be assessed. Both, the pre- and the post-measurements will take place within two weeks prior to starting or after completing the intervention.

DETAILED DESCRIPTION:
BACKGROUND:

Simultaneous motor-cognitive training interventions are considered promising to prevent the decline in cognitive functioning in older adults with mild neurocognitive disorder (mNCD) and can be highly motivating when applied in form of exergames. To ameliorate the effectiveness of exergaming, the neurobiological mechanisms as well as the most effective components for exergame interventions remain to be established. Besides establishing the most effective components [i.e., qualitative (e.g., type and content of training) and quantitative (e.g., frequency, intensity/complexity, session duration, intervention dose and adaptation over time) exercise and training variables] of exergames for cognition, it is crucial to also account for the users' perspective when designing and developing novel exergames or training concepts.

On this basis, a novel exergame-based training concept (called the 'Brain-IT' exergame-based training concept) was developed specifically for older adults with mNCD with the aim to halt and/or reduce cognitive decline and improve quality of life in older adults with mNCD. This exergame-based training concept has been developed on basis of a structured, iterative, and evidence-based approach based on a theoretical framework - The 'Multidisciplinary Iterative Design of Exergames (MIDE): A Framework for Supporting the Design, Development, and Evaluation of Exergames for Health'. The 'Brain-IT' exergame-based training concept represents a guideline for applying exergame-based motor-cognitive training by standardizing the training characteristics (e.g. training frequency, duration), as well as the structure and content of the training, whereas the exergame device and the games used within each of the defined neurocognitive domains can be replaced at will by alternative exergames. In this study, our training concept is implemented using the 'Senso (Flex)' (Dividat AG, Schindellegi, Switzerland), because this training device is already widely used for motor-cognitive training within geriatric populations, physiotherapies or in rehabilitation in Switzerland and was found to be suitable to implement our training concept. A step-by-step explanation of our methodological approach including the basis for the decision for the design of the exergame-based training concept as well as the complete 'Brain-IT' exergame-based training concept with sufficient details to allow full replication has been published as a methodological paper (doi: 10.3389/fnagi.2021.734012). The 'Brain-IT' exergame-based training concept has already been tested in a pilot randomized controlled trial and has shown good results in feasibility (i.e. recruitment, adherence, compliance, attrition), usability (i.e. system usability), and acceptance (i.e. enjoyment, training motivation and perceived usefulness) (unpublished work; NCT04996654). Based on the findings of this study, some minor modifications were incorporated to optimize the training concept so that it can be applied in a larger sample of patients to be evaluated on its effectiveness to halt and/or reduce cognitive decline and improve quality of life in older adults with mNCD.

OBJECTIVES & HYPOTHESES:

This study explores the effectiveness of the 'Brain-IT' training to improve global cognitive func-tioning in older adults with mNCD. With this, we aim to get a sufficiently precise estimate of the treatment effect to minimize the sample needed for a future full-scale RCT.

Null Hypothesis (H0): In older adults with mNCD, the addition of the 'Brain-IT' training to usual care has no significant effect on global cognitive functioning compared to usual care.

Alternative Hypothesis (HA): In older adults with mNCD, the addition of the 'Brain-IT' training to usual care results in differing effects on global cognitive functioning compared to usual care.

As secondary objectives, the effects of the 'Brain-IT' training on: (1) domain-specific cognitive functioning (i.e. learning and memory, complex attention, executive function, and visuospatial skills), (2) brain structure and function, (3) spatiotemporal parameters of gait, (4) IADL and (5) psychosocial factors (i.e. QoL, and levels of depression, anxiety, stress), and (6) cardiac vagal modulation (i.e. resting vagally-mediated heart rate variability (vm-HRV)) in older adults with mNCD as compared to usual care will be explored. Brain structure and function will be evaluated to explore possible underlying neural changes of the training in relation to adaptations in cognitive performance. For the remaining outcomes, the following hypotheses were formulated:

Null Hypothesis (H0): In older adults with mNCD, the addition of the 'Brain-IT' training to usual care has no significant effect on (1) domain-specific cognitive functioning, (3) spatiotemporal parameters of gait, (4) IADL and (5) psychosocial factors (i.e. QoL, and levels of depression, anxiety, stress), and (6) cardiac vagal modulation (resting vm-HRV) com-pared to usual care.

Alternative Hypothesis (HA): In older adults with mNCD, the addition the 'Brain-IT' training to usual care results in differing effects on (1) domain-specific cogni-tive functioning, (3) spatiotemporal parameters of gait, (4) IADL, (5) psychosocial factors (i.e. QoL, and levels of depression, anxiety, stress), and (6) cardiac vagal modulation (resting vm-HRV) com-pared to usual care.

METHODS:

A two-arm, parallel-group, single-blinded (i.e. outcome evaluator of pre- and post-measurements blinded to group allocation) randomized controlled trial with an allocation ration of 1 : 1 (i.e. intervention : control) including 34 - 40 older adults with mNCD will be conducted between May 2022 and December 2023.

After recruitment, interested subjects will be screened on eligibility between May 2022 and September 2023. All potential subjects will be fully informed about the study procedures by providing verbal explanations and an information sheet. Expected effects, benefits and risks of the study will be explained by the investigators, who will also be available to answer open questions and clarify uncertain-ties of participants. It will further be verified, that withdrawal is permitted at any time during the study without having to give a reason. After sufficient time for considerations (i.e. at least 24 h after handing out the study information sheet, but on average around two weeks), suitable patients willing to take part in the study will provide written informed consent in a second in-person meeting with the study team at the interested persons' home or at one of the study centres, depending on their preferences. If eligible patients decline to participate in the study, all data researched by their doctors or therapists and submitted to the study team will be permanently deleted. After providing written informed consent, the participants will be fully screened on eligibility, and the third study appointment (pre-measurements) will be scheduled. For participants recruited in the area of Zurich, the pre-measurements will take place at ETH Hönggerberg (Robert-Gnehm-Platz 1, CH-8093 Zurich). For participants recruited in the area of St.Gallen, the pre-measurements will take place at Eastern Switzerland University of Applied Sciences (Vadianstrasse 29, CH-9000 St.Gallen). The measurements will take approximately 60 - 90 min. For all participants who have no contraindications to MRI, an additional appointment to conduct the MRI scan will be scheduled. The MRI scan will take place at University Hospital Zurich (Rämistrasse 100, CH-8006 Zurich) and will take approximately one hour (including preparation). After completing the pre-measurements, participants will be randomly allocated to the intervention group (i.e. 'exergame group') or control group (i.e. 'usual care'). All participants will be instructed about their respective intervention procedures. For participants in the exergame group, the device will be installed at their homes, they will get a safety instruction and will be familiarized with the exergame training system 'Senso Flex', and the study intervention will be started according to the newly developed 'Brain-IT' exergame-based training concept (see section 'Intervention'). After completing the twelve-week intervention period, post-measurements (POST) will be performed for both groups. Both, the pre- and the post-measurements will take place and within two weeks prior to starting or after completing the intervention. No compensation will be granted to the participants, but detailed feedback on individual performance as well as the study outcomes in general will be provided at the end of the trial if desired.

ELIGIBILITY:
INCLUSION CRITERIA:

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* (1 = mNCD) clinical diagnosis of 'Mild Neurocognitive Disorder' according to the International Classification of Diseases 11th Revision (ICD-XI) or the Diagnostic and statistical manual of mental disorders (DSM-5®)) OR (2 = sMCI) patients screened for mild cognitive impairment (sMCI) according to the following criteria: (a) informant (i.e. healthcare professionals)-based suspicion of MCI confirmed by (b) an objective screening of MCI based on the German Version of the Quick Mild Cognitive Impairment Screen with (b1) a recommended cut-off score for cognitive impairment (MCI or dementia) of < 62/100 (doi: 10.3233/JAD-161204), while (b2) not falling below the cut-off score for dementia (i.e. < 45/100 (doi: 10.3233/JAD-161204)).
* German speaking
* able to stand at least for 10 min without assistance

EXCLUSION CRITERIA:

The presence of any of the following exclusion criteria will lead to exclusion of the participants:

* mobility impairments (i.e. gait, balance) that prevent experiment participation
* presence of additional, clinically relevant (i.e. acute and/or symptomatic) neurological disorders (i.e. epilepsy, stroke, multiple sclerosis, Parkinson's disease, brain tumors, or traumatic disorders of the nervous system)
* presence of any other unstable or uncontrolled diseases

Additional exclusion criteria will comprise of Covid-19 specific exclusion criteria (according to the Federal Office of Public Health). In case of Covid-19 specific exclusion criteria, participation in the study will only be allowed in case the treating physician provided written informed consent to allow participation in this study despite the presence of Covid-19 specific exclusion criteria. These Covid-19 specific exclusion criteria will include:

* high blood pressure (self-reported; systolic ≥ 140 mmHg and/or Diastolic ≥ 90 mmHg)
* Chronic respiratory condition
* uncontrolled type 2 Diabetes
* Condition or therapy that weakens the immune system
* unstable Cardiovascular Disease
* Cancer (present and/or under treatment)
* Serious obesity (BMI ≥ 40 kg/m2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Changes in Global Cognition | Both, the pre- and the post-measurements of the primary outcome measurement will take place within two weeks prior to starting or after completing the intervention.
  The German Version of the Quick Mild Cognitive Impairment Screen (Qmci) will be used to assess the overall level of cognitive functioning of the study population (doi: 10.1007/978-3-319-44775-9_12). Although being a screening instrument, the Qmci was shown to be equally sensitive with similar responsiveness to change over time as compared to the ADAS-Cog (which is considered the gold standard for assessing the efficacy of antidementia treatments) (doi: 10.3233/JAD-170991 and 10.3233/JAD-170991). The Qmci can be completed within 3 - 5 minutes and is scored as a point rate out of a maximum score of 100. It comprises six subtests: orientation (10 points), registration (5 points), clock drawing (15 points), delayed recall (20 points), verbal fluency (20 points), and logical memory (30 points). The Qmci will be administered according to the guidelines provided by O'Caoimh and Molloy in 2017 (doi: 10.1007/978-3-319-44775-9_12).

SECONDARY OUTCOMES:
Changes in Learning and Memory - Part 1 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Learning and memory will be assessed using the German version of the subtests 'logical memory' of the Wechsler Memory Scale-Revised (WMS-R-LM). The WMS-IV-LM is a measure of auditory verbal contextual learning and memory and has demonstrated excellent reliability and validity. The validated Older Adults battery (for ages 65 or older) of the German version of the WMS-IV-LM will be used for all participants. The test will be instructed, conducted and evaluated according to the standardized administration and scoring manual. During the 20 - 30 minutes retention phase, unrelated assessment (e.g. gait analysis, questionnaires) will be performed that to not interfere with memory.
Changes in Learning and Memory - Part 2 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Learning and memory will be assessed using a computerized version of the Digit Span Forward test (PEBL Digit Span Forward (PEBL-DSF)). The PEBL-DSF test will be used to assess immediate recall. It will be executed using the PEBL Test battery software (Version 2.1 (2); with default settings). Participants will have to remember and repeat digit sequences that are presented on the screen. Span length will cover two to a maximum of eight digits. For each digit span, two trials will be presented prior to increasing sequence length (in case at least one of the two trials was completed correctly). For every correct replication of a digit sequence, one point will be scored, summing up to a total point score. Additionally, the length of the longest correctly repeated digit sequence will be recorded as the maximum span. Instructions will be presented on the screen and will be explained verbally to each participant before starting the test.
Changes in Complex Attention - Part 1 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using a computerized version of the Trail Making Test - Part A (PEBL-TMT-A). The TMT-A is valid and reliable neuropsychological tests to assess psychomotor processing speed and visuoperceptual abilities. A computerized version of the of TMT-A (PEBL Test battery software (Version 2.1 (2); with default settings) will be used in this study. Participants will be instructed verbally and a short practice session will be conducted before starting the test. Completion time will be limited to 300 seconds. Completion times [s] (including the time for correction of errors) and number of errors will be measured.
Changes in Complex Attention - Part 2 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using the subtests 'Go-NoGo' of the Test of Attentional Performance (TAP Go-NoGo). The test of attentional performance (TAP; TAP Version 2.3.1, PSYTEST, Psychologische Testsysteme, Herzogenrath, Germany) is a valid and reliable computerized test battery to assess various attentional and executive functions. The TAP Go-NoGo will be used to assess selective attention and inhibition. The test form '1 of 2' will be instructed, conducted and evaluated according to the standardized protocol of the manufacturer. Median reaction times [ms] and number of errors [] will be measured.
Changes in Executive Function - Part 1 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  To measure planning ability, the HOTAP-A will be used. A set of photo cards containing actions typical for everyday life (e.g. making coffee, washing clothes, shopping) will be presented. The participants are verbally instructed to sort photo cards on which individual sub-steps of these typical everyday actions are depicted. The test will be instructed, conducted and evaluated according to the standardized protocol of the manufacturer. The outcome variable will be a combi score that is calculated by the sum of points divided by the time needed to arrange the cards.
Changes in Executive Function - Part 2 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  The PEBL Digit Span Backward (PEBL-DSB) [106-108] test will be used to assess working memory capacity. It will be instructed, administered, and scored identical to the PEBL-DSF (Outcome 3), but participants will have to remember and repeat digit sequences in reverse order.
Changes in Executive Function - Part 3 | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Complex attention will be assessed using a computerized version of the Trail Making Test - Part B (PEBL-TMT-B). The TMT-B is valid and reliable neuropsychological tests to assess cognitive flexibility. It consists of 25 randomly allocated circles distributed over a sheet of paper. A computerized version of the of the TMT-A (PEBL Test battery software (Version 2.1 (2); with default settings) will be used in this study. It will be instructed, administered, and scored identical to the PEBL-TMT-A (Outcome 4).
Changes in Visuospatial Skills | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Visuo-spatial functions will be tested with a computerized version of the classic Shepard and Metzler's mental rotation task [124]. The PEBL-Mental Rotation Task (PEBL-MRT) will be executed using the PEBL Test battery software (Version 2.1 (2); with default settings). Instructions will be presented on the screen and will be explained verbally to each participant before starting the task. Pairs of differently rotated two-dimensional polygons will be presented simultaneously on the screen. Participants will need to decide as quickly as possible whether the two presented objects are identical (i.e. pressing <Lshift> on the keyboard) or different (i.e. pressing <Rshift> on the keyboard). Median reaction time of correct answered trials [s] as well as performance (number of correct answered trials) will be measured as indicator for mental rotation ability. Trials with reaction times of less than 0.2 seconds or greater than 13 seconds will be excluded from data analysis.
Changes in Brain Structure and Function - Part 1 (Grey Matter Volumes) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Brain structure and function will be assessed by magnetic resonance imaging (MRI) using a 3.0 Tesla Philips whole-body scanner in all patients who have no contraindications to MRI to investigate more closely the underlying neural changes responsible for adaptations in cognitive performance. In Part 1, a 3D isotropic T1-weighted (T1w) scan (duration = 6.5 min) for assessing fine anatomical detail and brain atrophy (voxel size = 1.0 x 1.0 x 1.0 mm^3) and an acceleration factor of 2 (TFE-Sense: 2) will be conducted. The grey matter volumes will be determined for the following key regions of interest (ROIs): total brain (i.e. the total brain volume without the ventricles (brainsegvolnotvent) from the aseg file was used), hippocampus, dorsolateral prefrontal cortex (dlPFC), prefrontal cortex (PFC), anterior cingulate cortex (ACC).
Changes in Brain Structure and Function - Part 2 (White Matter Volumes) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Brain structure and function will be assessed by magnetic resonance imaging (MRI) using a 3.0 Tesla Philips whole-body scanner in all patients who have no contraindications to MRI to investigate more closely the underlying neural changes responsible for adaptations in cognitive performance. In Part 1, a 3D isotropic T1-weighted (T1w) scan (duration = 6.5 min) for assessing fine anatomical detail and brain atrophy (voxel size = 1.0 x 1.0 x 1.0 mm^3) and an acceleration factor of 2 (TFE-Sense: 2) will be conducted. The white matter volumes will be determined for the following key ROIs: total brain (i.e. the total brain volume without the ventricles (brainsegvolnotvent) from the aseg file was used), hippocampus, dorsolateral prefrontal cortex (dlPFC), prefrontal cortex (PFC), anterior cingulate cortex (ACC).
Changes in Brain Structure and Function - Part 3 (Mean diffusivity) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Brain structure and function will be assessed by magnetic resonance imaging (MRI) using a 3.0 Tesla Philips whole-body scanner in all patients who have no contraindications to MRI to investigate more closely the underlying neural changes responsible for adaptations in cognitive performance. In Part 2, diffusion tensor imaging (DTI, duration = 6 min) for the assessment of white matter microstructural integrity and connectivity, with resolution 2.0 x 2.0 x 2.0 mm^3, a minimum of 30 uniformly distributed directions with b = 1000 s/mm2, (EPI-Sense 2-32 directions; we use the vendor-provided directions set), and an acceleration factor of 2 will be conducted. Mean diffusivity will be calculated for parahippocampal white matter and the posterior cingulum, that were defined as key ROIs for this study.
Changes in Brain Structure and Function - Part 4 (Fractional Anisotropy) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Brain structure and function will be assessed by magnetic resonance imaging (MRI) using a 3.0 Tesla Philips whole-body scanner in all patients who have no contraindications to MRI to investigate more closely the underlying neural changes responsible for adaptations in cognitive performance. In Part 2, diffusion tensor imaging (DTI, duration = 6 min) for the assessment of white matter microstructural integrity and connectivity, with resolution 2.0 x 2.0 x 2.0 mm^3, a minimum of 30 uniformly distributed directions with b = 1000 s/mm2, (EPI-Sense 2-32 directions; we use the vendor-provided directions set), and an acceleration factor of 2 will be conducted. Fractional anisotropy will be calculated for parahippocampal white matter and the posterior cingulum, that were defined as key ROIs for this study.
Changes in Brain Structure and Function - Part 5 (Functional Connectivity Maps at rest) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Brain structure and function will be assessed by magnetic resonance imaging (MRI) using a 3.0 Tesla Philips whole-body scanner in all patients who have no contraindications to MRI to investigate more closely the underlying neural changes responsible for adaptations in cognitive performance. In Part 3, a task-free, eyes open (resting state) fMRI (duration = 9 min) for the assessment of functional networks and pathways using a T*2-weighted blood oxygen level-dependent (BOLD)-sensitive sequence, with resolution of 3.5 x 3.5 x 3.5 mm^3, TR = 2110 msec, and 300 volumes over time will be conducted. Individual functional connectivity maps for the hippocampal seed will be generated based on correlations between the mean signal time course within each seed region and the following selected key ROIs: precuneus/posterior cingulate cortex, medial prefrontal cortex, medial temporal lobe, angular gyrus, lateral temporal cortex and medial, lateral and inferior parietal cortex.
Changes in Brain Structure and Function - Part 6 (Functional Connectivity Maps during an episodic memory-task) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Brain structure and function will be assessed by magnetic resonance imaging (MRI) using a 3.0 Tesla Philips whole-body scanner in all patients who have no contraindications to MRI to investigate more closely the underlying neural changes responsible for adaptations in cognitive performance. In Part 4, a task-based (event-related) fMRI measured with an episodic memory task (face-occupation matching task) for the assessment of functional networks and pathways using a T*2-weighted blood oxygen level-dependent (BOLD)-sensitive sequence, with resolution of 3.5 x 3.5 x 3.5 mm^3, TR = 2110 msec, and 300 volumes over time will be conducted. Data will be analysed as described in 'Changes in Brain Structure and Function - Part 3'.
Changes in Spatiotemporal Gait Parameters - Part 1 (single-task gait speed at preferred walking speed) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be gait speed [m/s].
Changes in Spatiotemporal Gait Parameters - Part 2 (stride duration) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be stride duration [ms].
Changes in Spatiotemporal Gait Parameters - Part 3 (stride length) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be stride length [cm].
Changes in Spatiotemporal Gait Parameters - Part 4 (stance phase duration) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be stance phase duration [ms].
Changes in Spatiotemporal Gait Parameters - Part 5 (swing time) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be swing time [ms].
Changes in Spatiotemporal Gait Parameters - Part 6 (single support time) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be single support time [ms].
Changes in Spatiotemporal Gait Parameters - Part 6 (double support time) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  These spatiotemporal parameters of gait will be assessed using the portable BTS G-WALK® (BTS Bioengineering S.p.A., Garbagnate Milanese, Italy) inertial sensor that will be attached with semi-elastic belt to the lower back of the participant. A gait-analysis protocol consisting of a figure-8 walking path (i.e. distance between cones approximately 8 m) will be applied. At least 50 consecutive gait cycles will need to be accomplished to ensure reliability of spatial and temporal parameters of gait variability. Therefore, participants will - depending on their walking speed and stride length - perform five to ten repetitions of the figure-8 walking path at preferred walking speed. Comparative quantitative reference values for healthy older adults are available. The outcome variable will be double support time [ms].
Changes in Instrumental Activities of Daily Living (IADL) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  IADL functioning will be assessed using the Amsterdam IADL Questionnaire short version German for Switzerland, which has demonstrated good psychometric properties. In addition, the original version of the Amsterdam IADL questionnaire was sensitive to longitudinal changes and has been recommended for its use in research settings. The closest informant (e.g., spouse, child or friend) will fill out the questionnaire twice (within two weeks before the study participant starts or completes the intervention). Every item is scored on a five-point Likert scale ('no difficulty' to 'unable to perform'). The scoring is based on item response theory (IRT) of scoring. The IRT latent trait levels are transformed to a T-score, with a range from 20 to 80, a mean of 50 and standard deviation of 10. A higher T-score indicates better functioning.
Changes in Psychosocial Factors - Part 1 (Quality of Life) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Quality of life will be evaluated in interview format using the Quality of Life-Alzheimer's Disease (QOL-AD) scale. The QOL-AD is a valid and reliable self-report 13-item scale assessing various domains of QOL of cognitively impaired patients. The German version of the QOL-AD scale will be used that has shown to have a high test-retest reliability and good construct validity. It will be administered and evaluated according to the standardized instructions. Comparable values for patients with mNCD are available.
Changes in Psychosocial Factors - Part 2 (Symptoms of Depression) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  Levels of depression, anxiety, and stress will be assessed using the short version of the Depression, Anxiety and Stress Scale-21 (DASS-21). The DASS-21 was shown to have a high reliability and exhibits good convergent and discriminant validity when compared with other validated measures of anxiety and depression across age-groups. The validated German version of the DASS-21 will be administered and scored according the guidelines and scoring template. Existing normative data of the three subscales are available and suggest cut-off scores of 10, 8, or 15 to indicate significant depression, anxiety, or stress, respectively.
Changes in vagally-mediated Heart Rate Variability (HRV) | Both, the pre- and the post-measurements of all secondary outcome measurements will take place within two weeks prior to starting or after completing the intervention.
  To determine changes in resting HRV, all participants will be instructed to sit in a comfortable position on a chair without speaking, both feet flat on the floor with knees at a 90° angle, hands on thighs, and eyes closed. The measurement (10 min acclimatization followed by 5 min resting measurement) will be performed in a quiet room with dimmed light and at room temperature, using the heart rate monitor (Polar M430) and sensor (Polar H10). Mainly vagal-mediated HRV indices (i.e. mean R-R time interval (mRR), root mean square of successive RR interval differences (RMSSD), the percentage of successive RR intervals that differ by more than 50 ms (pNN50), the absolute power of the high-frequency band, the relative power of HF (in normal units), the Poincaré plot standard deviation perpendicular to the line of identity (SD1), and the parasympathetic nervous system tone index (PNS-Index) will be calculated using Kubios HRV Premium.

CONTACTS AND LOCATIONS:
Overall Officials: Eling D de Bruin, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Manser P, de Bruin ED. Making the Best Out of IT: Design and Development of Exergames for Older Adults With Mild Neurocognitive Disorder - A Methodological Paper. Front Aging Neurosci. 2021 Dec 9;13:734012. doi: 10.3389/fnagi.2021.734012. eCollection 2021. PMID 34955806
- [Result] Manser P, de Bruin ED. "Brain-IT": Exergame training with biofeedback breathing in neurocognitive disorders. Alzheimers Dement. 2024 Jul;20(7):4747-4764. doi: 10.1002/alz.13913. Epub 2024 May 29. PMID 38809948
- [Derived] Manser P, Michels L, Schmidt A, Barinka F, de Bruin ED. Effectiveness of an Individualized Exergame-Based Motor-Cognitive Training Concept Targeted to Improve Cognitive Functioning in Older Adults With Mild Neurocognitive Disorder: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 6;12:e41173. doi: 10.2196/41173. PMID 36745483